CLINICAL TRIAL: NCT05839210
Title: Lifestyle Intervention of Food and Exercise for Lymphoma Survivors (LIFE - L)
Brief Title: Lifestyle Intervention of Food and Exercise for Lymphoma Survivors
Acronym: LIFE-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Tracy E Crane, PhD, RDN, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20221298
Record Dates: First submitted 2023-03-31; First posted 2023-05-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Mediterranean Diet; Exercise Program
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LIFE-L Group (Experimental): Participants already undergoing chemotherapy treatment as per standard of care for 6 cycles will meet weekly via phone for 30-45 minutes with a health coach that will provide education on a Mediterranean diet and an exercise program.
  Interventions: Behavioral: LIFE-L Mediterranean Diet; Behavioral: LIFE-L Home-Based Exercise Program; Behavioral: Supportive Materials
- Control Group (Other): Participants in this group already undergoing 6 cycles of chemotherapy will receive study materials and two 30-45 minutes health coaching sessions four weeks post- intervention.
  Interventions: Behavioral: Supportive Materials

INTERVENTIONS:
Behavioral: LIFE-L Mediterranean Diet — Mediterranean Diet will include goals of: 4+ vegetable servings (2-4 cups) daily, 2+ fruit servings (1.5-2 cups) daily, 2+ whole grain servings daily, 1+ legume serving daily, 1+ serving nuts and seeds daily, and seafood 2 times per week. Limit or avoid highly processed foods, sugar-sweetened beverages and foods, processed meats, red meat, and alcohol.
  Arms: LIFE-L Group
Behavioral: LIFE-L Home-Based Exercise Program — The Home-Based Exercise Program will include goals of: 150+ minutes moderate or 75+ minutes vigorous exercise per week, completed in sessions of at least 10-minute duration, including daily aerobic exercise plus two resistance-based exercise sessions per week.
  Arms: LIFE-L Group
Behavioral: Supportive Materials — Participants will receive an informational study notebook, an exercise reference poster and videos, a Fitbit, and three stretch bands of different intensities. Participants will also receive supportive and informational text messages or emails three (3) times per week during the study; participants can opt-out of these messages.
  Participants will be requested to utilize the Fitbit app to track exercise sessions, as well as the MyFitnessPal app to track their diet. Support to set up apps will be provided by research staff. For participants who choose not to use the app, a laminated diet and exercise tracking sheet with dry erase marker will be provided, and participants will be advised to send a picture of their completed tracking sheet by text message to research staff each week.

SUMMARY:
The purpose of this study is to investigate if a mediterranean diet and exercise program for Lymphoma patients during chemotherapy can improve treatment completion and reduce treatment-related side effects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Any sex/gender
3. Able to provide consent
4. Able to read or understand English or Spanish
5. Diagnosis of untreated Non-Hodgkin or Hodgkin lymphoma, requiring at least 6 cycles of chemotherapy, being treated with one of the following therapies at discretion of PIs:

   1. R-CHOP or R-CHOP-like regimen
   2. BR
   3. BV-AVD or ABVD or checkpoint inhibitor+AVD
6. ECOG Performance Status grade of <2

   a. PI approval needed if ECOG = 2
7. Approval from treating oncologist, confirmed via email or in writing
8. Delivery of chemotherapy treatments at one of the following institutions:

   1. Sylvester Comprehensive Cancer Center (including satellite/network sites)
   2. University of Miami Hospital/UHealth Tower
9. Internet access on a smart phone, tablet, or computer
10. Willing to be randomized to a Mediterranean diet/home-based physical activity intervention or waitlist-control group.

Exclusion Criteria:

1. Individuals younger than 18 years of age
2. Unable to provide consent
3. Unable to read or understand English or Spanish
4. Any contraindication for diet change or exercising as determined by physician
5. Currently following a vegan or ketogenic diet, or consuming more than 5 servings of fruit and vegetables per day for the prior month
6. Engaging in >150 minutes of moderate to vigorous physical activity on average per week for the prior month
7. History of dementia or major psychiatric disease
8. History of recent (≤1 yr) stroke, myocardial infarction or congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Survivors who participate | Up to 12 months
  Percentage of survivors who agree to participate out of the total number of participants recruited will be assessed using a threshold of greater than or equal to (>=) 50-percent.
Percentage of Participants Completing Intervention Sessions | Up to 26 weeks (Post-Intervention)
  Percentage of intervention session completion at the end of treatment will be assessed, using a threshold of greater than or equal to (>=) 80-percent.
Change in percentage of participant satisfaction | 4 weeks (post-intervention), up to 30 weeks
  The change in percentage of participant satisfaction rate at the end of study participation will be assessed, using a threshold of greater than or equal to (>=) 80-percent. Participant satisfaction will be assessed via exit interviews.

SECONDARY OUTCOMES:
Average Relative Dose Intensity (RDI) | Up to 30 weeks
  RDI will be assessed using a threshold of greater than or equal to (>=) 80-percent.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy E Crane, Phd, RDN, Principal Investigator — University of Miami; Craig Moskowitz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No